CLINICAL TRIAL: NCT05365698
Title: A Quantitative Evaluation of the Community Health and Nutrition (CHN) Program in Jordan
Brief Title: Supporting Optimal Infant, Young Child and Maternal Nutrition and Health in Jordan: An Evaluation of the CHN Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Shibani Ghosh, Research Associate Professor, Tufts University
Other Study IDs: 00001816
Record Dates: First submitted 2022-04-25; First posted 2022-05-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Evaluations
MeSH Terms: interventions — Public Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort I: randomly assigned 12 health facilities (treatment/intervention group) that will have access to CHN program components
  Interventions: Behavioral: Community Health and Nutrition Program
- Cohort II: randomly assigned 12 health facilities that will serve as a control for the first year of the program implementation and then transition into the intervention/treatment group
  Interventions: Behavioral: Community Health and Nutrition Program

INTERVENTIONS:
Behavioral: Community Health and Nutrition Program — The "Community Health and Nutrition" supported by the United States Agency for International Development (USAID) will be implemented by an international NGO, FHI 360. The goal of the Community Health and Nutrition (CHN) program is to improve the nutritional status of pregnant and lactating women (PLW) and children under the age of two years in the target areas of the Hashemite Kingdom of Jordan. The program will fulfill this goal by implementing activities to support improvements in IYCF practices, increase adoption of optimal family planning practices and maternal, infant and young child nutrition (MIYCN) practices, and by improving health care provider support for proper IYCF practices and use of modern contraceptive methods.

SUMMARY:
The purpose of the comprehensive evaluation is to assess USAID supported Community Health and Nutrition (CHN) program's ability to effect change, the comprehensive evaluation will assess the effectiveness of CHN in influencing the knowledge, attitudes, practices, motivation, and support of health care providers, as well as the behavior change in pregnant and lactating women of reproductive age and their infants/young children thus supporting optimal maternal, infant and young child nutrition and health.

DETAILED DESCRIPTION:
Breastfeeding (BF) plays an important foundation for a healthy and well-developed child, and complementary feeding (CF) builds upon this foundation. Appropriate timing and introduction of high-quality complementary foods are key to sound infant, young child feeding (IYCF) practices. There is compelling evidence that BF and CF are crucial for the growth and development of a child, and in preventing malnutrition. Given this context, the USAID-supported "Community Health and Nutrition" (CHN) is being implemented in three governorates (Amman, Karak, Zarqa) of Jordan to improve the nutritional status of pregnant and lactating women (PLW) and children under the age of two years. The program will fulfill this goal by implementing activities to support improvement in IYCF practices, increase adoption of optimal family planning practices and maternal, infant, and young child nutrition (MIYCN) practices, and by improving health care provider support for proper IYCF practices and use of modern contraceptives methods (MCMs).

The purpose of the comprehensive evaluation is to assess USAID supported Community Health and Nutrition (CHN) program's ability to effect change. The evaluation will assess the effectiveness of CHN in influencing the knowledge, attitudes, practices, motivation, and support of health care providers, as well as the behavior change in pregnant and lactating women of reproductive age and their infants/young children thus supporting optimal maternal, infant and young child nutrition and health.

The study will utilize a cluster-randomized stratified stepped wedge design with two steps and two strata (cohort I and cohort 2). The stepped wedge study design is a staggered rollout design in which treatments are introduced to clusters at different time points. This design is particularly well suited for evaluating large-scale programs, like CHN, that roll out the intervention across clusters in phases. The use of strata (stratification) ensures representation of both regional and facility-level differences across the two cohorts.

The investigators will conduct 4 repeat annual cross-sectional surveys on women of reproductive age who are pregnant or are lactating and have a child under 2 years of age. Women will be recruited in the facilities and data will be collected at 12-month intervals. They will also conduct 3 repeat annual cross-sectional surveys on service providers (health care providers and community health agents) who work at these health facilities and within districts that are targets of the CHN program.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and Lactating women with child under 2 years:

Currently a beneficiary of CHN (except at baseline, prior to CHN implementation) Pregnant or lactating women (18-49 years) with children under the age of two years Willing to participate in the study and able to provide informed consent Currently lives within the study area

* Service providers:

Currently working in a CHN accredited social franchise facility Currently working in a maternal and child health department and actively providing services to PLWs Willing to participate in the study Received training from CHN on integrated maternal and child nutrition and healthcare services

Exclusion Criteria:

* Pregnant and Lactating Women with child under 2 years Not willing to participate or provide informed consent Not living in the study area
* Service providers No specific exclusion criteria

Ages: 18 Years to 49 Years | Sex: Female
Age Groups: Adult
Study Population: Jordanian Pregnant women and lactating women between 18 to 49 years who have a child under two years of age and are visiting a participating health facility targeted by the CHN program will be eligible to participate in the comprehensive evaluation.
  Healthcare providers and community based agents from the participating health facility targeted by the CHN program will be eligible to participate in the service providers' evaluation
Sampling Method: Probability Sample
Enrollment: 1145 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Diet Diversity in Pregnant and Lactating women | 2024
  Percentage of pregnant and lactating women meeting the minimum dietary diversity for women metric (MDDW)
Early initiation of breastfeeding | 2024
  Percentage of women who initiate breastfeeding within the first hour of birth
Exclusive breastfeeding | 2024
  Percentage of women who exclusively breastfeed their infants from birth to 6 months of age
Median duration of exclusive breastfeeding | 2024
  Increased median duration of exclusive breastfeeding (months) in infants aged 0-6 months
Improved nutritionally adequate diet and safe complementary feeding in infants and young children 6-23 months | 2021
  Percentage of children aged 6-23 months achieving a minimum acceptable diet (MAD)
Improved post party family planning | 2024
  Percentage of women using modern contraceptive improved postpartum practice on the use of modern contraceptive methods

CONTACTS AND LOCATIONS:
Overall Officials: Shibani Ghosh, PhD, Principal Investigator — Tufts University
Locations (1):
- Mindset, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Researchers outside of Tufts requesting access to the study data will be required to enter into a data-sharing agreement (modeled after examples such as the AHRQ National Inpatient Sample http://www.ahcpr.gov/data/hcup/datause.htm.) This agreement will: (i) require requesters to protect participants' privacy and data confidentiality (and restrictions against attempting to identify study participants), (ii) prohibit the recipient from transferring the data to other users; (iii) require destruction of the data after the planned analyses are completed; (iv) require that the data be used for research purposes only; (v) requires proper acknowledgment of the data resource; and (vi) require IRB approval from the requester's institution.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: publicly accessible in 2027-28
Access Criteria: Anyone who wishes to have access to the de-identified dataset for any research purpose will have access to the data. Data will be publicly available in the United States Agency for International Development's (USAID) Development Data Library (DDL), and Tufts Research Data Management platform.URLs will be added later once the data is successfully uploaded and data-sharing URLs have been generated.